CLINICAL TRIAL: NCT04313179
Title: Music Therapy as an Adjuvant Therapy for Pain Management During Heel Prick Procedures in Term Neonates.
Brief Title: Music Therapy for Pain Management for Minor Procedures in Neonates.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic prevented further enrollment. Interim analysis showed adequate power achieved.
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Pratiba Ankola, MD, Neonatologist, New York City Health and Hospitals Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB#18-026
Record Dates: First submitted 2020-03-09; First posted 2020-03-18 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Pain
Keywords: Neonatal pain; Music therapy
MeSH Terms: conditions — Pain | interventions — Music Therapy; Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music group (Experimental): "Deep Sleep" music track from "Bedtime Mozart: Classical Lullabies for Babies", played through smart phone speakers, at maximum sound up to 45 dB, starting 20 minutes before the heel prick procedure, continuing through the procedure and for 5 minutes after the procedure. Also given 0.5 ml of 24% Sucrose given 2 minutes prior to heel prick procedure for baseline pain relief.
  Interventions: Other: Music therapy; Other: Sucrose
- Placebo group (Placebo Comparator): 0.5 ml of 24% Sucrose given 2 minutes prior to heel prick procedure. No music played.
  Interventions: Other: Sucrose

INTERVENTIONS:
Other: Music therapy — Mozart lullaby music
  Arms: Music group
Other: Sucrose — 0.5 ml of 24% Sucrose

SUMMARY:
The aim of this study is to assess the effectiveness and safety of music therapy as adjuvant therapy for pain management in newborns undergoing minor painful procedures. It is a prospective study and we plan to enroll 200 healthy full term newborns undergoing minor procedures (heel pricks). They will be randomly assigned to either control or music group. Those in music group will receive recorded Mozart lullaby music. Pain will be assessed using NIPS (Neonatal Infant Pain Scale) scoring tool. The potential benefit of the study would be identifying music a safe and efficient adjuvant therapy for pain management in newborns.

DETAILED DESCRIPTION:
This randomized, controlled, double blinded, clinical trial will include full term neonates undergoing painful minor procedures (heel pricks) in the Nursery unit of Lincoln Medical and Mental Health Center.

One of the investigators involved in the study will obtain consent from the legal guardian and enroll the participants. All infants, regardless of the group that they are assigned, will receive similar standard non-pharmacologic method of pain relief which is 0.5 ml of 24% Sucrose, 2 minutes before undergoing heel prick. Pacifiers will be avoided to avoid potential confounding.

Subjects will be randomized into two different groups. Group A, music intervention group and group B, control group. In the music intervention group, a recorded instrumental lullaby music track called "Deep Sleep" from "Bedtime Mozart: Classical Lullabies for Babies", will be played for the neonates through smart phone speakers (maximum sound up to 60 A dB), starting 20 minutes before the heel prick, continuing through the procedure and for 5 minutes after the procedure. This music track has been selected based on previous research studies that showed effectiveness in neonatal pain management.

An investigator involved in the study will place the baby in a bassinet in a quite, dim lighted room. He/She will play the music for those babies in the music group and will NOT assess the NIPS. Another investigator wearing active noise cancelling Bluetooth headphones (for blinding) will enter the room at 5 minutes prior to the procedure and assess the NIPS at appropriate intervals: 5 minutes prior and at 1-minute interval during and after the procedure for 5 minutes. NIPS will be compared using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* >37 weeks gestation babies

Exclusion Criteria:

* <37 weeks gestation babies
* Major congenital anomalies
* Failed hearing screen

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Reduction in NIPS scoring by 20% | 5 minutes post procedure
  A score greater than 3 indicates pain, maximum score is 7 and minimum is 0

CONTACTS AND LOCATIONS:
Overall Officials: Prathiba Ankola, MD, Principal Investigator — Lincoln Medical Center
Locations (1):
- Lincoln Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Standley J. Music therapy research in the NICU: an updated meta-analysis. Neonatal Netw. 2012 Sep-Oct;31(5):311-6. doi: 10.1891/0730-0832.31.5.311. PMID 22908052
- [Background] Bieleninik L, Ghetti C, Gold C. Music Therapy for Preterm Infants and Their Parents: A Meta-analysis. Pediatrics. 2016 Sep;138(3):e20160971. doi: 10.1542/peds.2016-0971. Epub 2016 Aug 25. PMID 27561729
- [Background] Shukla VV, Bansal S, Nimbalkar A, Chapla A, Phatak A, Patel D, Nimbalkar S. Pain Control Interventions in Preterm Neonates: A Randomized Controlled Trial. Indian Pediatr. 2018 Apr 15;55(4):292-296. Epub 2018 Feb 9. PMID 29428919